CLINICAL TRIAL: NCT06881615
Title: A Randomized Clinical Trial Comparing Hydraulic Cements in Partial Pulpotomy in a Madrid Population: Impact of Clinical and Procedural Variables on Treatment Outcomes
Brief Title: Hydraulic Cements in Partial Pulpotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Ruth Perez Alfayate, full professor, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-305; CI 2023-305 (Other: UEMadrid)
Record Dates: First submitted 2025-02-26; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-01

CONDITIONS: Pulpitis; Caries Active
Keywords: partial pulpotomy; hydraulic cements; hemostasis
MeSH Terms: conditions — Pulpitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- MTA (Experimental): MTA PLACEMENT FOR PP
  Interventions: Device: MTA PLACEMENT FOR PP
- PUTTY (Experimental): PUTTY PLACEMENT FOR PP
  Interventions: Device: PUTTY PLACEMENT FOR PP

INTERVENTIONS:
Device: MTA PLACEMENT FOR PP — MTA PLACEMENT FOR PP
  Arms: MTA
Device: PUTTY PLACEMENT FOR PP — PUTTY PLACEMENT FOR PP
  Arms: PUTTY

SUMMARY:
This study is a randomized clinical trial that compares two types of hydraulic cements used in partial pulpotomy procedures for permanent teeth affected by deep decay and pulp inflammation. The purpose of the study is to determine which cement results in better treatment outcomes, such as preserving tooth vitality, reducing pain, and promoting healing. All patients receive a standardized treatment procedure and are then randomly assigned to one of the two cement groups. Key factors such as the time required to achieve hemostasis, the size of the pulp exposure, and other clinical variables are evaluated. Patients are followed up at 15 days and at 1, 3, 6, and 12 months after treatment to assess their clinical and radiographic outcomes. The results of this study will help improve treatment protocols and guide health care providers in selecting the most effective materials for partial pulpotomy.

DETAILED DESCRIPTION:
Study design and ethics This prospective single-arm randomized clinical trial followed the Preferred Reporting Items for Randomized Trials in Endodontics (PRIRATE) guidelines. After approval from the Institutional Investigation and Ethical Committee (CI: 2023-305 ) the research was conducted in the Department of Endodontics of the University . All participating patients were thoroughly informed about the advantages and disadvantages of opting for partial pulpotomy, as well as the differences and implications of choosing this treatment option over conventional endodontics. Furthermore, all patients signed an informed consent form, acknowledging the alternatives and associated risks. Only those patients who provided informed consent for the proposed treatment were included in the final analysis Sample size The sample size was determined using the conventional formula for estimating a single proportion. Assuming an anticipated success rate of 90% for the Vital Pulp Therapy procedure, a 95% confidence level (Z = 1.96) and an allowable margin of error of 7% were considered appropriate. The margin of error was set at 7% to balance statistical precision with clinical feasibility, acknowledging that in the context of vital pulp therapy, such a margin provides a reliable estimate of treatment success while accommodating practical limitations in patient recruitment and follow-up. Accordingly, the calculated minimum sample size was 71 cases.

Participant recruitment

From December 2022 to December 2023, patients presenting to the Department of Endodontics at the University were screened for eligibility. Inclusion criteria comprised patients diagnosed with initial, mild, moderate, or severe pulpitis according to the Wolters et al. (2017) classification, aged between 18 and 88 years, and having a non-contributory medical history. Furthermore, only permanent teeth affected by caries and exhibiting a proximity to the pulp-assessed via periapical and bitewing radiographs-with a distance ranging from 0 to 1.5 mm were selected. In addition, selected teeth were required to have fully formed apices, a periapical index score of ≤2, no tenderness on percussion, and probing pocket depths and mobility within normal limits. Exclusion criteria were defined as follows: patients diagnosed with pulp necrosis according to the American Association of Endodontists (AAE) guidelines; patients who declined vital pulp therapy as a treatment option; and patients with systemic conditions that could affect treatment outcomes. Additionally, teeth were excluded if they exhibited immature roots; if no pulp exposure occurred despite complete caries excavation; if bleeding after pulpal amputation could not be controlled within the prescribed time (10 minutes); if the pulp chamber was exposed to the oral environment; if insufficient bleeding was observed after pulp exposure-indicating necrotic or partially necrotic pulp; or if there was evidence of pathological root resorption, fracture or calcification. A total of 97 cases were initially analyzed, and after excluding 26 cases due to patient refusal of VPT, the predetermined sample size of 71 cases was reached. Enrollment was subsequently discontinued, as this number met the sample size requirements established by our statistical calculation. This approach ensured that the study maintained adequate power while preserving sample homogeneity, with all patients being treated by a single operator to guarantee procedural standardization.

Pulpal Diagnosis Pulpal diagnosis was established via a comprehensive clinical evaluation, emphasizing patient-reported symptoms. Cold thermal sensitivity was assessed using cotton pellets moistened with a cold spray Endo Frost Roeko (Coltene, Altstätten, Switzerland). The thermal response was quantified in two dimensions: intensity and duration. Intensity was rated on a scale from 0 to 10, where 0 denotes no pain, 1-3 indicate mild pain, 4-6 indicate moderate pain, and 7-10 indicate severe pain. Duration was evaluated on a scale from 1 to 4, with a score of 1 corresponding to 1-10 seconds, 2 to 11-20 seconds, 3 to 21 seconds up to 1 minute, and 4 to more than 1 minute. To assess and classify the patient's preoperative pain, the Numeric Rating Scale was employed. Other diagnostic tests included digital palpation, percussion with a mirror handle, periodontal probing using a CP-12 probe (Hu-Friedy), and transillumination to detect fractures.

In addition, radiographic assessments were conducted using periapical radiographs with a positioning device and bitewing radiographs, thereby ensuring full visualization of the tooth structure and at least 2 mm of the surrounding periapical tissue.

Clinical procedure The entire clinical procedure for each participant was performed by a single, experienced endodontist following a standardized protocol and under strict aseptic conditions. Local anesthesia was administered using 4% articaine with 1:200,000 epinephrine (Dermogen Farma S.A. Madrid, Spain), employing an infiltrative technique for the maxilla and a nerve block for the mandible, approximately 10-15 minutes prior to the procedure to ensure optimal pulpal anesthesia. Once anesthesia was confirmed, isolation was achieved using a rubber dam (Nic Tone, Bucharest, Romania) and appropriate clamp (Hu-Friedy, Chicago, United States). The rubber dam and tooth surface were then disinfected using cotton pellets saturated with 5.25% sodium hypochlorite (masterful formula). Following preparation of the operative field, any pre-existing restorations, carious lesions, and infected dentin were removed using a high-speed turbine and a contra-angle handpiece, with sterile high- and low-speed burs of various sizes under water coolant (Komet, Lemgo, Germany). Caries excavation was performed using a peripheral-to-central approach, addressing the outermost areas first before proceeding to the carious tissue adjacent to the pulp chamber. If necessary, proximal wall reconstruction was performed using a sectional matrix (Composi-tight 3D sectional matrix by Garrison Dental Solutions, Michigan, United States) and composite resin (Composite Estelite sigma quick, Tokuyama Dental Corporation, Tokyo, Japan). Upon pulp exposure, the cavity was irrigated with 1.5 mL of 2.5% sodium hypochlorite (masterful formula). Using a new sterile high-speed round diamond bur (Komet, Lemgo, Germany), inflamed pulpal tissue was removed to a depth of 2-3 mm (partial pulpotomy). Hemostasis was confirmed by applying gentle pressure with a sterile cotton pellet soaked in 2.5% sodium hypochlorite for 2 to 10 minutes. The exposed pulp was irrigated with EDTA, followed by saline solution, and subsequently dried using sterile cotton pellets. If bleeding control was not achieved, an additional 1 mm of pulpal tissue was removed using the same bur previously employed. The hemostasis procedure was then repeated by applying pressure with sterile cotton pellets soaked in sodium hypochlorite. This process was reiterated until complete bleeding control was obtained. If complete pulpotomy were required, that case would be excluded from the study and the treatment protocol would be modified accordingly. The time required to achieve hemostasis was measured using a chronometer, starting from the moment of pulp exposure until complete control of bleeding was achieved. The size of the pulpal exposure was measured using a CP-15 probe (CP-15 periodontal probe, Hu-Friedy Chicago, United States), recording the largest dimension of the exposed area. In cases of circular exposures, the diameter was measured, while for irregularly shaped exposures, the greatest width was recorded. If multiple exposures occurred in the same tooth, both the number and cumulative size of the exposures were documented by summing the diameters of each exposure. Subsequently, a computer-based randomization algorithm (REDCap's randomization module, Research Randomizer, Randomization.com) was employed to assign patients to the respective hydraulic cement treatment groups: MTA Angelus (Angelus Indústria de Productos Odontológicos, Londrina, Brazil) or TotalFill BC RRM Fast Set Putty (FKG Dentaire, Le Crêt-du-Locle, Switzerland). The cements were then prepared according to the manufacturer's instructions. A 2-3 mm layer of the selected material was applied to the cavity using a sterile ball spatula to ensure proper placement. Following cement application, an initial setting time of 15 minutes was observed, verified visually under magnification (Flexion Basic, CJ-Optik, Aßlar, Germany) and assessed using a sterile probe (CP-15 periodontal probe, Hu-Friedy Chicago, United States). Once the material began to harden, a light-curable resin-based liner (Fuji I, GC, Tokyo, Japan) was applied over the cement and polymerized for 20 seconds. The procedure was completed with definitive restoration using composite resin (Composite Estelite sigma quick, Tokuyama Dental Corporation, Tokyo, Japan).

Evaluation criteria All recruited participants who underwent the assigned pulpotomy procedures were instructed to return at 15 days post- intervention for pain assessment and at 1, 3, 6 and 12 months for clinical and radiographic evaluations, to be carried out by an investigator blinded to study groups. Participants were also advised to report earlier if any issues arose in relation to the treated tooth. Clinical and radiographic outcomes were considered the primary outcome measures, whereas pain assessment was considered the secondary outcome measure. This standardized follow-up protocol ensured that each patient was evaluated at uniform intervals, thereby facilitating reliable outcome comparisons.

Clinical and radiographic success Cases were classified as successful only when they satisfied both clinical and radiographic criteria. Clinical success was defined by the complete absence of discomfort or spontaneous pain in the treated tooth, beyond the immediate postoperative period. In addition, cases were deemed clinically successful if they exhibited no tenderness on percussion or palpation, no sinus tract formation, no soft tissue swelling, and no complaints of heightened sensitivity to thermal stimuli. The clinical evaluation also encompassed an assessment of periodontal status, restoration integrity, and pulp sensibility via the cold thermal test. Radiographic evaluation was independently performed by two experienced endodontists, with cases achieving a Periapical Index (PAI) score of ≤2 and demonstrating no evidence of furcal radiolucency or internal/external resorption being classified as radiographically successful. In all cases classified as failures, root canal treatment was performed to manage the patient's symptoms.

Data Collection and Recording During the procedure, systematic data collection was performed and recorded in an Excel spreadsheet. Variables were organized into columns, while individual cases were documented in rows. The following parameters were recorded and described in Table 1.

Confidentiality and Data Management To ensure patient confidentiality, data were stored using patient record numbers, with no reference to patient names. Additionally, a parallel Word document contained a summary of each case. Informed consent forms were signed by both the patient and the clinician and securely stored in the clinic

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with initial, mild, moderate, or severe pulpitis according to the Wolters et al. (2017) classification (Wolters et al., 2017),
* aged between 18 and 88 years
* having a non-contributory medical history.
* only permanent teeth affected by caries and exhibiting a proximity to the pulp-assessed via periapical and bitewing radiographs-with a distance ranging from 0 to 1.5 mm
* required to have fully formed apices,
* a periapical index score of ≤2,
* no tenderness on percussion
* probing pocket depths and mobility within normal limits.

Exclusion Criteria:

* patients diagnosed with pulp necrosis according to the American Association of Endodontists (AAE) guidelines("AAE Consensus Conference Recommended Diagnostic Terminology," 2009);
* patients who declined vital pulp therapy as a treatment option;
* patients with systemic conditions that could affect treatment outcomes.
* teeth were excluded if they exhibited immature roots;
* if no pulp exposure occurred despite complete caries excavation;
* if bleeding after pulpal amputation could not be controlled within the prescribed time (10 minutes)(Taha et al., 2017)

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — male and female
Enrollment: 71 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Clinical Success at 15 days | From enrollment to the end of treatment at 2 weeks
  Clinical success is defined as the absence of pain, absence of tenderness to percussion, and no sinus tract formation.
Number of Participants with Clinical Success at 1,3,6 months | From enrollment to the end of treatment at 1, 3, 6 months
  Clinical success is defined as the absence of pain, absence of tenderness to percussion, and no sinus tract formation.
Radiographic success | From enrollment to the end of treatment at 1, 3, 6, 12 months
  Number of Participants with Radiographic Success Based on Periapical Index (PAI) at 12 Months. Radiographic success is defined as a Periapical Index (PAI) score ≤ 2, evaluated by two independent endodontists.
Number of Participants with Clinical Success at 12 Months | participants enrolled from end of the treatment to 12 months
  Clinical success is defined as the absence of pain, absence of tenderness to percussion, and no sinus tract formation.
Mean Pain Score at 15 Days, 1,3,6 and 12 months Using the Numeric Rating Scale (NRS) | 15 days, 1 month, 3 months, 6 months and 12 months post-intervention
  Postoperative pain is assessed using the Numeric Rating Scale (NRS) from 0 to 10, where higher scores indicate greater pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Odontologica Universitaria Universidad Europea de Madrid, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
IF ANY RESEARCHER IS INTERESTED ON ANY INFORMATION OF THE STUDY WE WILL BE GIVING IT BY EMAIL CONTACT